CLINICAL TRIAL: NCT01526954
Title: A Prospective, Randomized, Controlled, Single-blind, Multicenter Clinical Trial Evaluating the Safety and Efficacy of the Cohera TissuGlu® Surgical Adhesive in the Management of Wound Drainage as Compared to the Standard of Care Closure Techniques Following Abdominoplasty
Brief Title: Cohera TissuGlu® Surgical Adhesive in the Management of Wound Drainage
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cohera Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO-100-0003
Record Dates: First submitted 2012-01-31; First posted 2012-02-06 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Abdominoplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- TissuGlu Surgical Adhesive (Experimental): Experimental Arm: standard of care plus TissuGlu Surgical Adhesive and no drains
  Interventions: Device: TissuGlu Surgical Adhesive
- Control- Standard of Care (No Intervention): Control Arm: standard of care plus drains and no TissuGlu Surgical Adhesive

INTERVENTIONS:
Device: TissuGlu Surgical Adhesive — TissuGlu Surgical Adhesive to be used prior to closure of the large tissue flap in abdominoplasty cases.
  Arms: TissuGlu Surgical Adhesive

SUMMARY:
This study is designed to evaluate the safety and efficacy of the device while reducing the amount of drainage from surgical wounds following large flap surgical procedures, in this case abdominoplasty, as compared to the standard of care (closure techniques). It is hypothesized that the use of the Cohera device will facilitate reduction or closure of dead space when applied to planar surfaces created during an abdominoplasty procedure.

DETAILED DESCRIPTION:
Background:

Fluid accumulation in dissected tissue planes has been a longstanding problem following surgical procedures. The common use of closed suction drains has been associated with infection risk, wound healing complications, additional scarring, and patient discomfort. Additionally, seroma formation after drain removal often requires invasive treatment. Therapies that can reduce fluid accumulation and decrease the need for drains will have a positive impact on surgical practice.

Objectives:

* To establish that the use of TissuGlu® Surgical Adhesive is a safe and effective alternative to drains (standard of care) for fluid management following abdominoplasty.
* To evaluate the impact of TissuGlu® Surgical Adhesive on post-operative invasive treatments, and seroma formation.
* To evaluate the impact of TissuGlu® Surgical Adhesive on post-operative subject satisfaction and quality of life.
* To document the type and duration of adverse events associated with TissuGlu® used during an abdominoplasty procedure as an alternative to drains.

Material and Methods:

A prospective randomized trial comparing standard wound closure technique with drains in 130 subjects (control group n=65) to standard wound closure techniques plus TissuGlu® and no drains (test group n=65) during Abdominoplasty.

For subjects randomized into the Test Group, TissuGlu® will be applied to one surface of the exposed tissue flap using the custom applicator during a standard abdominoplasty procedure followed by normal wound closure (suturing technique) without drain placement. The applicator device will deliver an array of drops spaced equidistant apart. The user may then reposition the device to the next area and repeat the application process. Each device will dispense approximately 5 ml of adhesive. It is expected that one 5 ml device will suffice for the average sized subject (400-500 sq cm tissue flap). The TissuGlu® is applied using the disposable applicator to the tissue surfaces to be adhered just prior to standard closure. The tissue is then approximated, and the wound is closed using standard suturing techniques. TissuGlu® will begin to cure upon exposure to moisture in the tissue. The cure process takes approximately 30-45 minutes.

Subjects that are randomized to the Control Group will undergo normal wound closure (suturing technique) and placement of two size 12 Blake drains.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* BMI ≤ 35;
* ≤ ASA2 - American Society of Anesthesiologists (ASA) Physical Classification System (2=patient with mild systemic disease);
* Be in good general health in the opinion of the Investigator with no conditions that would significantly impact wound healing as determined by medical history and review of recent concomitant medications;
* Be scheduled for at least one full thickness surgical incision of at least 20cm in length as part of elective abdominoplasty.
* Be willing to follow instructions for incision care, wound exudates volume measurements, and diary completion as instructed by the investigator, and follow guidelines related to resumption of daily activities;
* Agree to return for all follow-up evaluations specified in this protocol
* Agree not to schedule any additional elective surgical procedures that involve an incision on the abdomen, until their participation in this study is complete; and
* Sign the informed consent

Exclusion Criteria:

* Exclusion Criteria:
* Pregnant or breastfeeding
* Previous abdominoplasty;
* Concurrent liposuction during procedure;
* Use of pain pumps;
* Have severe co-morbid conditions (e.g., heart disease);
* Known medical condition that results in compromised blood supply to tissues;
* Any condition known to effect wound healing, such as collagen vascular disease;
* Are currently a smoker or have smoked within 30 days of prescreening as determined by nicotine test;
* Be known to have a blood clotting disorder and/or be willing to discontinue anti-coagulation therapy - including aspirin;
* Diagnosis of diabetes with current medical treatment;
* Be receiving antibiotic therapy for pre-existing condition or infection;
* Have known personal or family history of keloid formation or hypertrophic scarring;
* Undergoing concurrent adjacent or congruent Liposuction procedures;
* Concurrent use of fibrin sealants or other internal wound care devices;
* Be currently taking systemic steroids or immunosuppressive agents;
* Concurrent hernia repair greater than 6 cm and/or requiring the use of mesh;
* Mini abdominoplasty (Abdominoplasty without umbilical transposition);
* Have known or suspected allergy or sensitivity to any test materials or reagents; and
* Be participating in any current clinical trial or have participated in any clinical trial within 30 days of enrollment in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Time to reach drain removal criteria. | Measured until drains are removed, up to 30 days post-op.
  Primary efficacy endpoint is time (days) to reach drain removal criteria of less than 30ml per 24hr period.